CLINICAL TRIAL: NCT00002106
Title: A Pilot Randomized, Double-Blind, Placebo-Controlled, Parallel Design, Multicenter Trial to Evaluate the Effect of Ranitidine on Immunologic Indicators in Asymptomatic HIV-1 Infected Subjects With a CD4 Cell Count Between 400-700 Cells/mm3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Model: Parallel | Purpose: Treatment
Other Study IDs: 135A; RAN-809
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1994-05

CONDITIONS: HIV Infections
Keywords: Ranitidine
MeSH Terms: conditions — HIV Infections | interventions — Ranitidine

INTERVENTIONS:
Drug: Ranitidine hydrochloride

SUMMARY:
To evaluate the effect of ranitidine on immunologic indicators in asymptomatic HIV-1 infected patients with CD4 counts of 400-700 cells/mm3.

DETAILED DESCRIPTION:
Patients are randomized to receive either ranitidine or matching placebo bid for 16 weeks, with follow-up every 4 weeks through week 20.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Asymptomatic HIV-1 infection.
* CD4 count of 400-700 cells/mm3.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Significant illness.
* Acute illness at randomization.
* Hemodialysis.

Prior Medication:

Excluded:

* Antiretroviral use within 60 days prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Pacific Oaks Med Group, Sherman Oaks, California
  - Community Research Initiative, Coral Gables, Florida
  - Duke Univ Med Ctr, Durham, North Carolina
  - Houston Clinical Research Network, Houston, Texas

REFERENCES:
- [Background] Bartlett JA, Berry PS, Bockmon KW, Stein A, Johnson J, Quinn JB, Weinhold KJ. A placebo controlled trial of ranitidine in HIV infection. Natl Conf Hum Retroviruses Relat Infect (2nd). 1995 Jan 29-Feb 2:149